CLINICAL TRIAL: NCT07217457
Title: Epidural Wave Form Analysis vs Fluoroscopic Guidance for Thoracic Epidural Placement
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Alexander T. Abess, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02002726
Record Dates: First submitted 2025-10-12; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Epidural Placement
Keywords: epidural waveform; fluoroscopic guidance; thoracic epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Cohort (Experimental): The primary objective of this study is to assess the accuracy with which epidural waveform analysis (EWA) can confirm epidural access in comparison to the gold standard of fluoroscopic confirmation (FC). Our hypothesis is that FC is superior to EWA. We will determine the Positive Predictive Value and Negative Predictive Value of EWA referenced to FC.Every participant enrolled in the study will be in the experimental arm and will undergo epidural waveform analysis and fluoroscopic confirmation of epidural access.
  Interventions: Diagnostic Test: Epidural Waveform Analysis

INTERVENTIONS:
Diagnostic Test: Epidural Waveform Analysis — All participants in this study will undergo epidural waveform analysis (pressure measurements) and fluoroscopic guidance of epidural placement. Epidural waveform analysis as method to determine epidural access will be compared to fluoroscopic confirmation.

SUMMARY:
The primary objective of this study is to compare the effectiveness of epidural waveform analysis (EWA) with fluoroscopic guidance for confirmation of successful epidural placement. In this study, participants will undergo both EWA and fluoroscopy. EWA involves measuring the pressure in the epidural space once accessed and determining whether or not a waveform that corresponds with the participant's heart rate is present. The pressure measuring apparatus is the same that is used for direct pressure monitoring elsewhere in the body (i.e. invasive arterial catheters or intracranial pressure monitoring).

DETAILED DESCRIPTION:
The primary objective of this study is to assess the accuracy with which epidural waveform analysis (EWA) can confirm epidural access in comparison to the gold standard of fluoroscopic confirmation (FC). Our hypothesis is that FC is superior to EWA. We will determine the Positive Predictive Value and Negative Predictive Value of EWA referenced to FC.

If EWA performs reasonably well compared to FC, then EWA could be used in settings where anesthesia providers do not have access to fluoroscopy or the expertise to perform fluoroscopic-guided thoracic epidurals. EWA uses clinically approved pressure transducers, which are used commonly to analyze other physiologic pressures (e.g. invasive hemodynamic monitoring and invasive intracranial pressure monitoring.) and could offer a low budget way to help reassure that placement of a needle is indeed epidural, and not in a different location.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing surgery at Dartmouth Hitchcock Medical Center
* Scheduled for planned (non-emergent, non-urgent) thoracic epidural placement as part of surgery and anesthesia
* English speaking
* Must have capacity for consent

Exclusion Criteria:

* Non-english speaking
* Incarceration
* Pregnant
* Minors (under age 18)
* Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value and Negative Predictive Value of epidural waveform analysis to predict epidural access compared with fluoroscopic guidance | Time of enrollment through completion of epidural placement. Epidural placement occurs on study day 1 and is generally completed within 2 hours of study enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Abess, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
Participant privacy considerations remain paramount. De-identified data could be shared at some point if deemed helpful by other researchers and if approved by our institution review board and privacy officers.

REFERENCES:
- [Background] Hong JH, Jung SW. Analysis of epidural waveform for cervical epidural steroid injections confirmed with fluoroscopy. Medicine (Baltimore). 2018 Mar;97(13):e0202. doi: 10.1097/MD.0000000000010202. PMID 29595657
- [Background] Arnuntasupakul V, Van Zundert TC, Vijitpavan A, Aliste J, Engsusophon P, Leurcharusmee P, Ah-Kye S, Finlayson RJ, Tran DQ. A Randomized Comparison Between Conventional and Waveform-Confirmed Loss of Resistance for Thoracic Epidural Blocks. Reg Anesth Pain Med. 2016 May-Jun;41(3):368-73. doi: 10.1097/AAP.0000000000000369. PMID 26894628